CLINICAL TRIAL: NCT00590850
Title: A Multicenter, Prospective, Randomized Trial of Non-Operative Versus Operative Treatment for High-Energy Midshaft Clavicle Fractures
Brief Title: Non-Operative Versus Operative Treatment for High-Energy Midshaft Clavicle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Orthopaedic Trauma Association (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHS-07-03-04
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-03

CONDITIONS: High Energy Midshaft Clavicle Fractures
MeSH Terms: interventions — Bone Plates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Closed (No Intervention): Closed Treatment
- ORIF (Active Comparator): Open Reduction and Internal Fixation (ORIF) with Plate and Screws
  Interventions: Procedure: ORIF with Plate and Screws
- Pin (Active Comparator): Pin Fixation
  Interventions: Procedure: Pin Fixation

INTERVENTIONS:
Procedure: ORIF with Plate and Screws — ORIF with plate and screws
  Arms: ORIF
Procedure: Pin Fixation — Clavicle fixation with clavicle pin
  Arms: Pin

SUMMARY:
Clavicle (collar bone) fractures account for about 33% of all fractures around the shoulder. Some surgeons suggest that surgical treatment is the best option, while others suggest that nonoperative care is the best treatment. There is no evidence to date that either option in superior. For this reason, we propose to conduct a prospective, randomized clinical trial of surgical versus non-surgical treatment of displaced high-energy clavicle fractures. This study will use both objective clinical and patient-based outcome measures. The purpose of this study is to see if there is a difference between clinical outcomes (healing rate, time to healing, time to return to work, Constant Score, complications), functional outcomes (DASH Score), and health related quality of life (SF-36) in nonoperative care and two types of surgical care for displaced fractures of the clavicular shaft in adults.

Included patients will be randomized into one of three groups: nonoperative care (Group N); surgical care using plates and screws (Group P); and surgical care using intramedullary pin put inside of the clavicle to stabilize it (Group I).

ELIGIBILITY:
Inclusion Criteria:

* ages of 18 and 85
* a midshaft clavicle fracture
* fracture displaced the width of the clavicle or shortened at least 1.5 cm
* less than 21 days since the injury

Exclusion Criteria:

* injury involving the lateral ligaments
* fracture involve the sternoclavicular joint
* Pathologic Fracture
* Open Fracture
* Fracture with neurovascular compromise
* Displaced fracture with impending skin compromise
* Medical comorbidities that preclude surgery
* Associated injuries to ipsilateral shoulder girdle
* severe cognitive disability or injury that may inhibit study form completion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2003-10; Primary Completion 2020-12 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Disability of Arm, Shoulder and Hand (DASH) scores | 1 year
  Disability of Arm, Shoulder and Hand (DASH) scores

SECONDARY OUTCOMES:
Reoperation rate | 1 year
  rate of reoperations between groups

CONTACTS AND LOCATIONS:
Overall Officials: Kyle J Jeray, MD, Principal Investigator — Greenville Hospital System
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeray KJ, Broderick JS, Mullis BH, Everhart J, Tanner SL, Snider BG; Southeastern Fracture Consortium. Multicenter, Prospective, Observational Study of Nonoperative Versus Operative Treatment for High-Energy Midshaft Clavicle Fractures. J Orthop Trauma. 2024 Jul 1;38(7):345-350. doi: 10.1097/BOT.0000000000002817. PMID 38837208